CLINICAL TRIAL: NCT05204953
Title: Mean Platelet Volume and Its Relation to Risk Stratification of Myelodysplastic Syndromes
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Consultant of Clinical Hematology, Assiut University
Other Study IDs: PVARMDS
Record Dates: First submitted 2022-01-09; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: patients diagnosed to have myelodysplastic syndrome
- 2: healthy control subjects

SUMMARY:
The myelodysplastic syndromes (MDS) are a group of myeloid neoplasms characterized by abnormal differentiation and maturation of myeloid cells, reduced bone marrow (BM) function, and a genetic instability with enhanced risk to transform to secondary acute myeloid leukemia, AML

DETAILED DESCRIPTION:
The diagnosis of MDS is an effort that requires clinicians and pathologists to work together. A patient's life, livelihood and outlook can be profoundly affected by the terms used by the treating physician. The typical presentation is unexplained anemia, leukopenia and/or thrombocytopenia, in an older patients (median age ≥ 70 years). However, thrombocytosis may be associated with the 5q-deletion syndrome or in selected patients with refractory anemia with ringed sideroblasts syndrome . The white count may be elevated in MDS / myeloproliferative disorder overlap syndromes particularly in chronic myelomonocytic leukemia, CMML.

MDS remains among the most challenging of the myeloid neoplasms to diagnose and classify, particularly in cases in which the blast percentage is not increased in the peripheral blood or bone marrow. Diagnostic problems can arise when the clinical and laboratory findings suggest MDS, but the morphologic findings are inconclusive; when there is secondary dysplasia caused by nutritional deficiencies, medications, toxins, growth factor therapy, inflammation or infection; or when marrow hypocellularity or myelofibrosis obscures the underlying disease process .

The prognosis of MDS is determined by several factors. Revised International Prognostic Scoring System (IPSS-R) for MDS divides patients into very low, low, intermediate, high and very high risk groups. Five factors (the percentage of bone marrow myeloblasts, the diagnostic cytogenetics, the hemoglobin level, the platelet count and the absolute neutrophilic count) are used to generate a prognostic score .

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed to have myelodysplastic syndromes

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed to have myelodysplastic syndromes
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
mean platelet volume | at diagnosis (baseline)

SECONDARY OUTCOMES:
risk stratification of MDS patients | at diagnosis (baseline)
relation of MPV to risk stratification | at diagnosis (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: youssreya A Ahmad, MD, Study Director — Assiut University; Ahmad F Thabet, MD, Study Director — Assiut University

REFERENCES:
- [Background] Tefferi A, Lim KH, Levine R. Mutation in TET2 in myeloid cancers. N Engl J Med. 2009 Sep 10;361(11):1117; author reply 1117-8. doi: 10.1056/NEJMc091348. No abstract available. PMID 19741235
- [Background] Greenberg PL, Attar E, Bennett JM, Bloomfield CD, De Castro CM, Deeg HJ, Foran JM, Gaensler K, Garcia-Manero G, Gore SD, Head D, Komrokji R, Maness LJ, Millenson M, Nimer SD, O'Donnell MR, Schroeder MA, Shami PJ, Stone RM, Thompson JE, Westervelt P; National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: myelodysplastic syndromes. J Natl Compr Canc Netw. 2011 Jan;9(1):30-56. doi: 10.6004/jnccn.2011.0005. PMID 21233243
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Background] Foran JM, Shammo JM. Clinical presentation, diagnosis, and prognosis of myelodysplastic syndromes. Am J Med. 2012 Jul;125(7 Suppl):S6-13. doi: 10.1016/j.amjmed.2012.04.015. PMID 22735753
- [Background] Johnston TC, Thompson RB, Baldwin TO. Nucleotide sequence of the luxB gene of Vibrio harveyi and the complete amino acid sequence of the beta subunit of bacterial luciferase. J Biol Chem. 1986 Apr 15;261(11):4805-11. PMID 3514602
- [Background] Mittelman M, Oster HS, Hoffman M, Neumann D. The lower risk MDS patient at risk of rapid progression. Leuk Res. 2010 Dec;34(12):1551-5. doi: 10.1016/j.leukres.2010.05.023. Epub 2010 Jun 22. PMID 20573398